CLINICAL TRIAL: NCT05676333
Title: Pilot Trial to Determine the Efficacy of Secukinumab in Active Non-segmental Vitiligo
Brief Title: Secukinumab in Active Non-segmental Vitiligo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/0237
Record Dates: First submitted 2016-10-06; First posted 2023-01-09 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Vitiligo; Secukinumab
Keywords: Vitiligo; Secukinumab
MeSH Terms: conditions — Vitiligo | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Secukinumab (Experimental)
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab

SUMMARY:
Vitiligo is an acquired autoimmune skin disorder which leads to cutaneous depigmentations. A lot of progress has been made to unravel the pathophysiology of vitiligo. Several independent studies confirmed the elevated values of IL-17 in the serum of vitiligo patients and higher IL-17 values have been linked to a higher affected body surface area and a longer disease duration. The study will be a pilot trial with secukinumab in patients with active, non-segmental vitiligo. All patients will receive the active compound (= no placebo arm) as the purpose of the study is to investigate the potential efficacy of secukinumab in vitiligo.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to extensive vitiligo
2. Vitiligo patients with active vitiligo.
3. Vitiligo on hands and/or face
4. Fitzpatrick skin type 3-6
5. High impact

Exclusion Criteria:

1. Active systemic infections during the 2 weeks prior to baseline (exception: common cold) or any infection that reoccurs on a regular basis.
2. Autoimmune diseases (except thyroid disease)
3. Use of immunosuppressive treatments
4. Pregnancy or breastfeeding
5. Mycobacterium tuberculosis infection as shown by positive Mantoux and/or Quantiferon test
6. Clinical important abnormalities in blood analysis before start
7. Use of any other investigational drug within 4 weeks prior to baseline or within a period of 5 half-lives of the investigational drug, whichever is langer (in order to assess properly the safety of secukinumab)
8. History of hypersensitivity to any of the studied drugs or to drugs of similar chemical classes including latex hypersensitivity
9. Important underlying medical conditions
10. Significant medical problems
11. Serum creatinine level exceeding 2.0 mg/dL (176.8 pmol/L) at screening.
12. Total white blood cell (WBC) count < 2500/pL, platelets < 100 000/pL, neutrophils < 1500/ML or hemoglobin < 8.5 g/dL, at screening.
13. Past medical history record of, or current infection with, human immunodeficiency virus (HIV), hepatitis B virus or hepatitis C virus prior to baseline.
14. History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years (except for skin Bowen's disease, or basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 12 weeks; carcinoma in situ of the cervix or noninvasive malignant colon polyps that have been removed).
15. Current severe progressive or uncontrolled disease which in the judgment of the Investigator renders the patient unsuitable for the study or puts the patiënt at increased risk (eg, myocardial infarction within 26 weeks prior to baseline).
16. Inability or unwillingness to undergo repeated venipuncture (eg, because of poor tolerability or lack of access to veins).
17. Any medical or psychiatric condition which, in the investigator's opinion, would preclude the patient from adhering to the protocol or completing the study per protocol.
18. History or evidence of ongoing alcohol or drug abuse, within the last 6 months prior to baseline.
19. Plans for administration of live vaccines during the study period or in the 6 weeks prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2017-12-16 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Repigmentation (percentage of repigmentation) | 9 months
  The efficacy of the treatment will be determined by measuring the diffference in the percentage of the affected body surface area compared to baseline. The percentage of the affected body surface area will be measured by standardized digital pictures using a validated scoring system (Vitiligo Extent Score plus; VESplus).

SECONDARY OUTCOMES:
Stabilisation of disease (percentage of affected body surface area) | 9 months
  The efficacy of the treatment will be determined by measuring the diffference in the percentage of the affected body surface area compared to baseline. The percentage of the affected body surface area will be measured by standardized digital pictures using a validated scoring system (Vitiligo Extent Score plus; VESplus).
Disease impact | 9 months
  Global impact score (0-10), where the higher the score the worse the outcome
Satisfaction with treatment | 9 months
  Global Satisfaction Score, where the higher the score the better the outcome

CONTACTS AND LOCATIONS:
Overall Officials: van Geel Nanja, MD, PhD, Principal Investigator — Department of Dermatology, Ghent University Hospital
Locations (1):
- Department of Dermatology, Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No